CLINICAL TRIAL: NCT04122638
Title: Prevalence of Sarcopenia and Sarcopenic Obesity in Community-dwelling Outpatient Older Adults
Brief Title: Prevalence of Sarcopenia and Sarcopenic Obesity in Older Adults
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Collaborators: Istanbul Medeniyet University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Filiz Demirdağ, Principal Investigator, Goztepe Training and Research Hospital
Other Study IDs: GoztepeTRH
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Sarcopenia; Sarcopenic Obesity; Osteopenia, Osteoporosis
Keywords: Older adults
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Syndromes such as sarcopenia, sarcopenic obesity and osteosarcopenic obesity are commonly seen in older adults. They result from the impairment of muscle, bone and adipose tissue. Thus, they lead to a decrease in quality of life and increase morbidity and mortality. The aim of this study is to report the prevalence of sarcopenia, sarcopenic obesity and osteosarcopenic obesity in community-dwelling outpatient older adults and to investigate the related factors.

ELIGIBILITY:
Inclusion Criteria:

* Being at the age of 65 or older
* Being able to complete 4-m walk test

Exclusion Criteria:

* <24 points on Mini-Mental State Examination
* 12 points or higher on Geriatric Depression Scale

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults
Sampling Method: Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Handgrip Strength | 10 minutes
  Handgrip strength measured by Takei© Hand Dynamometer
Muscle mass | 5 minutes
  Using Bioimpedance analysis (BİA) technique with TANITA© TBF 300
Bone density | 30 minutes
  T score evaluation using Dual-energy X-ray absorptiometry (DEXA)
Percentage of body fat | 5 minutes
  Using Bioimpedance analysis (BİA) technique with TANITA© TBF 300

SECONDARY OUTCOMES:
Gait speed | 3 minutes
  4-m usual walking speed test
Physical Activity | 5-10 minutes
  Using Rapid Assessment of Physical Activity (RAPA)
Nutritional Status | 10 minutes
  Assessed with Mini-Nutritional Assessment (MNA)
Activities of Daily Living | 10 minutes
  Activities of daily living assessed with Katz Index of Independence in Activities of Daily Living
Instrumental Activities of Daily Living | 10 minutes
  Instrumental activities of daily living assessed with Lawton -Brody Instrumental Activities of Daily Living Scale
Depression | 10 minutes
  Assessed with The Geriatric Depression Scale- Short Form
Mini-Mental State Examination | 10-15 minutes
  Mini-Mental State Examination
Blood Sample Analysis | 5 minutes
  A blood sample analysis including parameters such as: wbc, hgb, htc, mcv ,plt, fasting blood sugar, urea, uric acid, creatin, AST, ALP, ALT, GGT, LDH, total colesterol, trigylicerid, LDL, HDL, NA, K, Mg, Ca, P, Albumin, protrombin time, CRP, B12, folate, iron, ferritin, PTH, vitamin-D, sedimentation, TSH, T4, insukin, HGBA1C, IHOMA-IR.
Comorbidities | 5 minutes
  Assessed with Charlson Comorbidity Index

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirdag F, Kolbasi EN, Aykut GB, Guler KY, Murat S, Ozturk GB, Oguz A. Nutritional status as a mediator between the age-related muscle loss and frailty in community-dwelling older adults. Arch Gerontol Geriatr. 2022 Jan-Feb;98:104569. doi: 10.1016/j.archger.2021.104569. Epub 2021 Nov 3. PMID 34768160